CLINICAL TRIAL: NCT05014035
Title: Feasibility of a Hybrid Delivery of Home-based Cluster Set Resistance Training in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ciaran Fairman, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00110261
Record Dates: First submitted 2021-07-30; First posted 2021-08-20 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer; Resistance Exercise
Keywords: Exercise; Physical Activity; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity; Lung Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental)
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — This is an 8-week exercise program, delivered using a hybrid approach of in-person, in-home supervised exercise, and virtual delivery of exercise via zoom. Individuals will participate in resistance exercise 3 days per week for 8 weeks.

SUMMARY:
Symptom burden remains a critical concern for individuals with non-small cell lung cancer (NSCLC) following the completion of treatment. Of those, symptom clusters such as dyspnea (shortness of breath) and fatigue, contribute to physical decline, reductions in quality of life, and a higher risk of comorbidities and mortality. It has been proposed that dyspnea is a primary limiter of exercise capacity in individuals with lung cancer, resulting in exercise avoidance and an accelerated physical decline. As such, specifically designing resistance exercise programs with cluster sets, to mitigate feelings of dyspnea and fatigue may result in improved exercise tolerance, resulting in the maintenance of physical function and quality of life.

The purpose of this project is to investigate the feasibility and preliminary efficacy of a hybrid-delivery of home-based cluster-set resistance exercise in individuals with NSCLC. Methods: Individuals with NSCLC (n=15), within 12-months of completion of treatment will be recruited to participate in this single arm feasibility trial. Participants will complete 8-weeks of home-based resistance training (RT) designed to target dyspnea and fatigue. The hybrid-delivery of the program will include supervised sessions in the participants home, and virtual supervision via video conferencing. The primary outcome of feasibility will be measured via recruitment rates, retention, acceptability and intervention fidelity. Exploratory outcomes (dyspnea, fatigue, quality of life, physical function and body composition) will be assessed pre- and post- intervention.

DETAILED DESCRIPTION:
Analysis plan. Descriptive statistics (percentages and means (with standard deviations)) will be used to report on feasibility outcomes (recruitment, retention, fidelity etc.). Unless explicitly stated, means and standard deviations will be reported for assessments of exploratory outcomes at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Completed definitive treatment for localized NSCLC (stages I-III)
* Has access to stable internet access for Zoom participation
* Willing to complete an 8-week, home-based intervention program that includes face-to-face and Zoom interaction.
* Willing to consider behavior change at this time.
* Able to speak and read English.
* Capable of informed consent
* Has obtained medical clearance from medical practitioner or medical team

Exclusion Criteria:

* Individuals with a known diagnosis of advanced lung cancer (stage IV; due to potential added burden) or diagnosis of small-cell lung cancer,
* Anyone for whom physical activity is not recommended.
* aren't comfortable having study staff visit their homes for exercise sessions
* have any neuromuscular, cardiovascular, or psychological condition precluding safe exercise;
* have participated in structured RE ≥2 times/week for the past 6 months;
* are unable to read/understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Recruitment | Through study completion, an average of 1 year
  The recruitment goal of n=15 is reached
Retention | Through study completion, an average of 1 year
  If ≥75% of the sample recruited to participate return for follow up testing
Intervention Fidelity | Through study completion, an average of 1 year
  Exercise fidelity will be reported using metrics previously outlines by Fairman et al (2019). Specifically, volume load will be calculated as a function of sets x reps for each exercise and summed to give total volume for each session. We will report the proportion of volume achieved relevant to what was prescribed to give a "relative-dose intensity" (RDI) for each person. RDI will then be averaged and used to determine fidelity to the RT intervention.

SECONDARY OUTCOMES:
Acceptability | At post intervention (8-weeks)
  10-item scale adapted from McDonnell et al (PMID: 33118443). Questions assessing the acceptability of the intervention will be scored on a 4-point Likert-Type scale from "Strongly disagree" to "Strongly Agree". Questions will ask about the utility of virtual exercise sessions, use of technology and level of tailoring the intervention
Dyspnea | Baseline and post intervention (8-weeks)
  Functional Assessment of Chronic Illness Therapy-Dyspnea (FACIT-D) 10-Item short form (parts 1 and 2). Part 1 assesses Dyspnea and Part 2 assesses dyspnea-associated functional limitations. Min score for each part: 0; max score for each part: 30. Higher scores indicate worse dyspnea/burden
Fatigue | Baseline and post intervention (8-weeks)
  Functional Assessment of Chronic Illness Therapy-Fatigue scale 13-item scale. Min score: 0 Max score: 52 Higher scores mean higher quality of life.
Lung Cancer Related Quality of Life | Baseline and post intervention (8-weeks)
  Functional Assessment of Cancer Therapy - Lung Cancer Subscale (LCS). Min score: 0; max score: 28. Higher scores indicate better quality of life.
Upper Body Muscular Strength | Baseline and post intervention (8-weeks)
  Chest Press five repetition maximum
Lower Body Muscular Strength | Baseline and post intervention (8-weeks)
  Leg Press five repetition maximum
Physical Function STS | Baseline and post intervention (8-weeks)
  5 times sit-to-stand (in seconds)
Physical Function 6MWT | Baseline and post intervention (8-weeks)
  6-minute Walk Test (distance in meters)
Fat Mass | Baseline and post intervention (8-weeks)
  Fat mass (kg) Dual Energy X-Ray Absorptiometry
Fat Free Mass | Baseline and post intervention (8-weeks)
  Fat Free Mass (kg) Dual Energy X-Ray Absorptiometry
Total Mass | Baseline and post intervention (8-weeks)
  Total Mass (kg) Dual Energy X-Ray Absorptiometry
Body Fat Percentage | Baseline and post intervention (8-weeks)
  Dual Energy X-Ray Absorptiometry
Appendicular Lean Mass | Baseline and post intervention (8-weeks)
  Sum of Arm and Leg Fat Free Mass
Bone Mineral Density | Baseline and post intervention (8-weeks)
  Total z-score Dual X-ray Absorptiometry
Acceptability | Post-Intervention (8-weeks)
  Qualitative interview with participants regarding the acceptability, likes, dislikes about the intervention and potential barriers for future participation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data and code for analyses will be made available as soon as possible with publication of the primary outcome paper. The dataset will include demographic information, and physiological and psychosocial measures outlined in the proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All de-identified data and code for analyses will be made available as soon as possible with publication of the primary outcome paper.
Access Criteria: We will make the de-identified data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.

REFERENCES:
- [Derived] Fairman CM, Owens OL, Kendall KL, Steele J, Schumpp AR, Latella C, Jones MT, Marcotte L, Dawson JM, Peddle-McIntyre CMJ, McDonnell KK. Hybrid delivery of cluster-set resistance training for individuals previously treated for lung cancer: the results of a single-arm feasibility trial. Pilot Feasibility Stud. 2023 Oct 17;9(1):177. doi: 10.1186/s40814-023-01405-z. PMID 37848969